CLINICAL TRIAL: NCT00440921
Title: Randomized Clinical Trial for Fibrin Sealant in Knee Surgery
Brief Title: Clinical Trial for Fibrin Sealant in Knee Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No agreement between investigator and sponsor
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: MDM (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RP06.008
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Total Knee-replacement; Total Hip-replacement
Keywords: fibrin sealnat; knee replacement; hip replacement; woud healing; blood loss; clinical trial; randomized
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Single donor Allogenous Fibrin Sealant

SUMMARY:
* Thermogenesis is a company that sells a machine for the production of fibrin sealant of single donor plasma, the CryoSeal Fibrin Sealant System (CS-1).
* Fibrin sealant consists of two components: cryoprecipitate and thrombin. Cryoprecipitate is the fraction of human plasma that contains concentrated coagulation factors, such as fibrinogen. Thrombin is an enzyme that facilitates the conversion of fibrinogen into fibrin, so that a clot will be formed.
* Fibrin sealant can be used in surgery to increase hemostasis in the wound after e.g. knee- or hip replacement, cosmetical surgery or partial liverresections.
* Until now, mainly autologous plasma was used to produce fibrin sealant with the CS-1. Within Sanquin there is a question whether fibrin sealant can be produced from the allogeneic quarantaine plasma that is in stock. Therefore in this study will be studied whether allogenous single donor fibrin sealant produced using the CS-1 is effective in wound healing and as consequence of this can be registered as a product of Sanquin. To answer these questions a national working party is formed, working party Fibrin Sealant.
* So far, three man personnel in Sanquin Blood Bank Nort East Region (SBNO) are certified by Thermogenesis to use the CS-1 for production of fibrin sealant and an in vitro validation has been performed.
* The next step will be a study for the in vivo effectiveness of fibrin sealant produced of single donor allogeneic quarantaine plasma using the CS-1. As control patients without fibrin sealant treatment will be studied. Two hospitals (Refaja Hospital in Stadskanaal and Wilhelmina hospital in Assen) are already interested in participating in this study. Probably, three more hospitals will participate.
* The use of fibrin sealant will be studied in a prospective randomized trial for patients undergoing knee and hip replacements.

DETAILED DESCRIPTION:
1. Introduction

   * Until now, mainly autologous plasma was used to produce fibrin sealant with the CS-1. Within Sanquin there is a question whether fibrin sealant can be produced from the allogeneic quarantaine plasma that is in stock. Therefore in this study will be studied whether allogenous single donor fibrin sealant produced using the CS-1 is effective in wound healing and as consequence of this can be registered as a product of Sanquin.
   * The use of fibrin sealant will be studied in a prospective randomized trial for patients undergoing knee and hip replacements.
2. Aim

   · To study the effectiveness of fibrin sealant produced of single donor allogeneic plasma when used intra-operatively after total knee or hip replacement.
   * Primairy endpoint: wound healing.
   * Secondary endpoints: total blood loss until 24h post-operative, amount of blood transfused, motion of the joint (knee) after surgery, amount of pain after surgery, use of antibiotics, wound infections, stay in hospital, adverse events, satisfaction with fibrin sealant as used by the physician.
3. Hypothesis

   * We hypothesize that use of fibrin sealant will have a positive effect on wound healing, will cause less blood loss, decreased use of antibiotics and and will cause that a decreased number of infections will be seen compared to patients who are not treated with fibrin sealant. Through this, hospital stay will probably be shortened for patients who are treated with fibrin sealant.
   * As a working hypothesis we assume a score for wound healing of at least 20% lower and at least 20% less blood loss for the fibrin sealant treated group.
4. Definitions

   · N/A
5. Ethical aspects 5.1 Admission of the Ethical Committee · For this study approval is asked from the ethical committee of each participating hospital.

   5.2 Admission of the patient

   · Each patient who potentially can be included will be asked with informed consent for admission and participation in the study.

   5.3 Confidentiality

   · Patients will be registered using a patient number, date of birth and study number and further will be anonimized.

   5.4 Input Data

   · Input of data will be done by the (senior) researcher O&O of SBNO. She/he will take confidentiality of the data into account.
6. Materials and collaborating departments

   * Orthopedic Surgery department of hospitals
   * Patient data (can be filled in on the forms in the appendix)
   * Fibrin Sealant data (can be filled in on the form in the appendix)
   * Department O&O of SBNO for analysis of data
   * SBNO for production and release of fibrin sealant
7. Patients 7.1 Inclusion

   * Age, minimum of 18 years
   * Gender, man or woman
   * Admission of the patient after informed consent 7.2 Exclusion
   * Liver failure
   * Congenital or acquired coagulation disorders
   * Thrombocytopenia, < 100 x10^9PLT/L 7.3 Number of patients
   * The number of patients needed in this study to indicate a statistical significantly difference can be calculated from a pilot study for wound healing in patients that have undergone knee- or hip replacement.
   * Knee replacement: For calculation of the number of patients we aim to see a significant difference of at least 20% better wound healing after use of fibrin sealant during surgery. From a pilot we observed for wound healing a score of 0.71±0.49. With the power at 80% and alpha at 0.05 we need 193 evaluable patients in both study group (fibrin sealant treated) and control group (non fibrin sealant treated).
   * Hip replacement: For calculation of the number of patients we aim to see a significant difference of at least 20% better wound healing after use of fibrin sealant during surgery. From a pilot we observed for wound healing a score of 1.58±0.79. With the power at 80% and alpha at 0.05 we need 96 evaluable patients in both study group (fibrin sealant treated) and control group (non fibrin sealant treated).
8. Adverse events

   * Each adverse event (AE) that occurs during of after the use of fibrin sealant will be noted on the form by the physician on duty.
   * An AE is any untoward medical occurrence in a patient ("patient" is defined as any subject who has been enrolled in the study as evidenced by the subject having signed informed consent) or any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease that occurs during the course of the clinical investigation. The AE may or may not be considered as related to the investigational drug or device. All AE's should be recorded in the patient's chart and graded mild, moderate, or severe. All AE's shall be handled to the hospital procedures in force and as soon as possible passed down to the study coordinators, in case of fatality at least within 24h.

     * Mild: Symptom barely noticeable to patient; does not influence performance or functioning. Prescription drugs not ordinarily needed for relief of symptom but may be given because of personality of patient.
     * Moderate: Symptom of sufficient severity to make patient uncomfortable; performance of daily activities influenced; patient is able to continue in study; treatment for symptom is needed.
     * Severe: Symptom causes severe discomfort, or may be of such severity that patient cannot perform daily routines, may cause cessation of treatment with fibrin sealant; or even may be fatal.
   * After complementary follow-up the physician on duty will conclude with notice of argumentation whether the AE:

     * is not caused by fibrin sealant
     * is possible, but not necessary caused by fibrin sealant (causes cannot be proven nor excluded)
     * is probably caused by fibrin sealant
     * is certainly caused by fibrin sealant
9. Procedure 9.1 Set up clinical trial

   * The study is a randomized prospective clinical trial.
   * Fibrin sealant treated patients will be compared with non fibrin sealant treated patients.
   * Patients included undergo total knee or hip replacement.
   * During participation of the patient, only the study coordinator of the hospital and the staff of the operation room know whether a patient is treated with fibrin sealant or not.
   * Nurses and patients can be informed at the end of participation of the patient (at discharge of the hospital).
   * Primairy endpoint is wound healing.
   * Secondary endpoints are total blood loss until 24h post-operative, amount of blood transfused, motion of the joint (knee) after surgery, amount of pain after surgery, use of antibiotics, wound infections, stay in hospital, adverse events, satisfaction with fibrin sealant as used by the physician.
   * Each group (fibrin sealant treated and non fibrin sealant treated) wil contain 193 patients for knee and 96 patients for hip surgery.

   9.2 Production and release of fibrin sealant

   · Fibrin sealant will be produced and released from SBNO according to the procedures in force.

   9.3 Controled treatment with fibrin sealant
   * Each patient who might be included (see 7.1 and 7.2) will be asked for admission to participate in this study by informed consent prior to surgery. Therefore a letter with information about this study will be given to each patient who might be included.
   * After admission an envelope will be openend by the study coordinator in the hospital in which a code is for treatment or no treatment with fibrin sealant. The study coordinator will tell the outcome only to the personel of the OR who need to know it for preparation and usage of the fibrin sealant. People from the operation room do not communicate this outcome to the nursery. Except for treatment with fibrin sealant there will be no difference in treatment of the patients.
   * Patient and nurses (when desired) will be informed about treatment with fibrin sealant or not when the patient leaves the hospital and is discharged from this study.
   * Prior to surgery a blood sample of the patient will be taken to determine the platelet count, hematocrit and hemoglobin.
   * Fibrin sealant, if used, will be assessed just before closing the wound. 9.4 Parameters
   * The following parameters of patients and surgery will be noted pre-operative by nurses (double blinded):

     * Birth date, gender
     * Weight, length
     * Platelet count, haemoglobin and hematocrit
     * Underlying diseases
     * Medication
     * Use of antibiotics
     * Pain (VASC) via standardized score: Score 0: no pain; 2: pain that can be neglected 4: uncomfortable pain; 6: painful, cannot be neglected; 8: very painful, patient cannot concentrate him/herself; 10: extreme painful, patient cannot do anything.
   * The following parameters of patients and surgery will be noted per-operative by staff of the operation room (single blinded):

     * Time points of start surgery, treatment with fibrin sealant and end of surgery
     * Hemostasis of fibrin sealant seen (yes or no), only for hip replacement, because it is hard to see this for knee replacement
     * Medication
     * Use of antibiotics
     * Number of transfusions (red cells, platelets and plasma)
     * Adverse events (severeness and relation to treatment with fibrin sealant)
     * Mobility of knee (only for knee replacement).
   * The following parameters of patients and surgery will be noted at 1h post-operative by staff of operation room (single blinded):

     * Blood loss via drain
     * Medication
     * Use of antibiotics
     * Number of transfusions (red cells, platelets and plasma)
     * Adverse events (severeness and relation to treatment with fibrin sealant)
     * Pain (VASC) at <1h after end of anaesthesia via standardized score (see above under parameters pre-operative).
   * The following parameters of patients and surgery will be noted >1h post-operative by the nurses (double blinded):

     * Wound healing including wound leakage and wound infection (via score form, see appendix) at time of wound treatment in case of heavy wound leakage (i.e. bandage need to be changed), at 3 days postoperatively and at discharge from hospital
     * Blood loss via drain at removing of the drain, mostly the next morning after surgery
     * Medication until discharge of hospital
     * Use of antibiotics until discharge from hospital
     * Number of transfusions (red cells, platelets and plasma) until discharge from hospital
     * Adverse events (severeness and relation to treatment with fibrin sealant) until discharge from hospital
     * Pain (VASC), at 3h post operative, at 21:00 h (day of surgery), at 8:00 h, 14:00 h and 21:00 h at day after surgery, at 8:00 h on the second day after surgery and at discharge from hospital as described above (under parameters pre-operative)
     * Mobility of knee at discharge from hospital. Also date at which 90° flexion is reached will be noted
     * Hospital stay after surgery in days
10. Analyzing and reporting of results 10.1 Analyzing results

    * Anonimized patient data will be put in and analyzed in an Excel file.
    * Results of knee and hip replacements will be analyzed and reported separately.
    * Via an unpaired t-test differences in primary and secondary endpoints between fibrin sealant treated and non fibrin sealant treated patients will be studied.
    * The Fisher's exact test will be used to determine the effect of use of fibrin sealant in wound leakage, wound infections and undesired events.
    * Of the results a report will be written. Also a report for data of each separate hospital will be written. Results about knee and hip replacements will described separately.
11. Time scheduling

    * The study will start in January 2007. After minimaal 193 evaluable patients per group for knee surgery (193 patients treated with fibrin sealant and 193 patients not treated with fibrin sealant) and minimal 96 evaluable patients per group for hip surgery (96 patients treated with fibrin sealant and 96 patients not treated with fibrin sealant) the study will be finished.
    * It is expected that this study will take about 1 year, in case 5 hospitals participate.
    * Only in case of serious reasons (e.g. severe adverse events) the study will be terminated early.

ELIGIBILITY:
Inclusion Criteria:

* Age, minimum of 18 years
* Gender, man or woman
* Admission of the patient after informed consent

Exclusion Criteria:

* Liver failure
* Congenital or acquired coagulation disorders
* Thrombocytopenia, < 100 x10^9 PLT/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
wound healing

SECONDARY OUTCOMES:
total blood loss until 24h post-operative
amount of blood transfused
motion of the joint (knee) after surgery
amount of pain after surgery
use of antibiotics
wound infections
stay in hospital
adverse events
satisfaction with fibrin sealant as used by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Coen van Delden, PhD, Study Chair — Sanquin Blood Bank North East Region